CLINICAL TRIAL: NCT00258141
Title: A Placebo-Controlled, Double-Blind, Cross-Over Study With Rupatadine 10 Mg in 30 Mosquito-Bite Allergic Adult Subjects
Brief Title: Study With Rupatadine in Mosquito-Bite Allergic Adult Subjects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: J. Uriach and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: DM03RUP/IV/05
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-11

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — rupatadine

INTERVENTIONS:
Drug: Rupatadine
Drug: Placebo

SUMMARY:
The study will find out how effective rupatadine is in the treatment of mosquito bite symptoms in adult patients allergic to mosquito bites.

DETAILED DESCRIPTION:
Mosquito-bite symptoms include wheals and pruritic bite papules. Oral antihistamines have shown to decrease whealing ang accompanying pruritus in placebo-controlled trials.

Subjects will be treated for 4 days, and exposed to experimental mosquito bite at day 3.

ELIGIBILITY:
Inclusion Criteria:

* Recent history of suffering from mosquito-bite reactions.
* At least 5 mm diameter mosquito-bite wheal from Aedes aegypti laboratory mosquitoes

Exclusion Criteria:

* Pregnancy or lactating females
* Oral antihistamines, corticosteroids or non-steroid anti-inflammatory drugs (NSAID) use within two weeks before the study.
* Severe or moderate systemic illness
* Allergy to rupatadine or other antihistamines
* Anaphylaxis from mosquito bites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

PRIMARY OUTCOMES:
Bite lesion size (squared mm)

SECONDARY OUTCOMES:
Pruritus on a Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Timo Reunala, Prof., Principal Investigator — Medical School, University of Tampere and Tampere University Hospital
Locations (2):
- Finland (2):
  - Ulappatorin Lääkäriasema, Espoo
  - Koskiklinikka, Tampere Lääkärikeskus, Tampere